CLINICAL TRIAL: NCT03338270
Title: Clinical Validation Study of a Novel Minute MRI Sequence
Brief Title: Clinical Validation Study of Multi-EPI Mix
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Anna Falk Delgado, Principal Investigator, Karolinska University Hospital
Other Study IDs: Neuroradiology Karolinska Uni.
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Brain Diseases
Keywords: MRI; Neuroradiology; minute-MRI; multi EPI-mix; Clinical Validation
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — MRI sequence without intravenous contrast

SUMMARY:
This study aims to assess the diagnostic validity of a new minute-MRI sequence for neuroradiological evaluation in comparison to conventional MRI.

DETAILED DESCRIPTION:
The study aims to assess the imaging quality with regards to artefacts and lesion conspicuity as well as its diagnostic potential in rendering a probable diagnosis. The primary study aim is to define the AUC for diagnostic performance of minute MRI compared to conventional MRI.

Included patients are those with suspiscion of cerebral pathology.

Study participancts are investigated at 3T.

ELIGIBILITY:
Inclusion Criteria:

- Neuroradiological MRI

Exclusion Criteria:

- Aborted exam

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neuroradiological indication for brain MRI
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic potential | At MRI scan. Diagnostic accuracy to categorize scan as normal or abnormal on a five point Likert scale compared to abnormal/normal conventional MRI.
  Diagnostic performance of lesion conspicuity of new MR sequence compared to conventional sequences

SECONDARY OUTCOMES:
Lesion location determination | At MRI scan
  Anatomical localization of abnormality
Lesion classification | At MRI scan
  Classification into disease categories
Imaging quality | At MRI scan
  Artefacts
Diagnostic imaging quality | At MRI scan
  Diagnostic imaging quality
Anatomical conspicuity | At MRI scan
  Specified anatomical structures
Multifocality | At MRI scan
  Determine multifocal lesion
Ability to rule out diseases | At MRI scan
  A list of diseases
Lesion description | At MRI scan
  For example effect on brain parenchyma and size
Diagnostic confidence | At MRI scan
  Scale
Brain coverage | At MRI scan
  Full or lower
Clinical diagnostic summay report | At MRI scan
  Text

CONTACTS AND LOCATIONS:
Overall Officials: Anna Falk Delgado, MD, PhD, Principal Investigator — Clinical Neuroscience
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Delgado AF, Kits A, Bystam J, Kaijser M, Skorpil M, Sprenger T, Skare S. Diagnostic performance of a new multicontrast one-minute full brain exam (EPIMix) in neuroradiology: A prospective study. J Magn Reson Imaging. 2019 Dec;50(6):1824-1833. doi: 10.1002/jmri.26742. Epub 2019 Apr 1. PMID 30932287